CLINICAL TRIAL: NCT03805022
Title: Phase III Trial Investigating the Potential Benefit of Intensified Peri-operative Chemotherapy With in High-risk CINSARC Patients With Resectable Soft-tissue SARComas
Brief Title: Benefit of Intensified Peri-operative Chemotherapy Within High-risk CINSARC Patients With Resectable Soft-tissue Sarcomas
Acronym: CIRSARC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: Novartis (Industry); Chugai Pharma France (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB 2017-04; 2018-000186-36 (EudraCT Number)
Record Dates: First submitted 2019-01-10; First posted 2019-01-15 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Non-metastatic Soft-tissue Sarcoma; Resectable
Keywords: Solid tumor; Phase III trial; Soft-tissue sarcoma; Resectable; Non-metastatic
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin; Ifosfamide; Dacarbazine

STUDY DESIGN:
Intervention Model Description: This is a multicenter trial with:
  * An open randomized two-arm phase III trial for high-risk CINSARC patients assessing whether the addition of 3 additional neo-adjuvant cycles of chemotherapy (doxorubicin based chemotherapy) to standard management (3 cycles of neoadjuvant anthracycline based chemotherapy + surgery +/- radiotherapy) improves the outcome of patients
  * a prospective cohort for low-risk CINSARC patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Control-Arm phase III high-risk CINSARC:
  Patients will be treated by doxorubicin (60 or 75mg/m² day or 20- or 25 mg/m² per day from day1 to day 3) + ifosfamide (7,5-9 g/m² over 3 days with mesna and G-CSF) or dacarbazine (100 mg/m² 1 day or 450 mg/m² 2 days) as per local practices of a 21-days cycle for up to 3 cycles in neoadjuvant setting Neoadjuvant chemotherapy will be followed by surgery. If indicated, radiotherapy could be prescribed at the discretion of the investigator (in neoadjuvant or adjuvant setting).
  Interventions: Drug: Doxorubicin; Drug: Ifosfamide or dacarbazine
- Arm B (Experimental): Experimental-Arm phase III high-risk CINSARC:
  Patients will be treated by doxorubicin (60 or 75mg/m² day or 20 or 25 mg/m² per day from day1 to day 3) + ifosfamide (7,5-9 g/m² over 3 days with mesna and G-CSF) or dacarbazine (100 mg/m² 1 day or 450 mg/m² 2 days) as per local practices of a 21-days cycle for up to 6 cycles in neoadjuvant setting Neoadjuvant chemotherapy will be followed by surgery. If indicated, radiotherapy could be prescribed at the discretion of the investigator (in neoadjuvant or adjuvant setting).
  Interventions: Drug: Doxorubicin; Drug: Ifosfamide or dacarbazine
- Prospective cohort (Experimental): Patients will be treated at the discretion of the investigator
  Interventions: Drug: At the discretion of the investigator

INTERVENTIONS:
Drug: Doxorubicin — A treatment cycle consists of 3 weeks. Doxorubicin will be administered from day 1 to day 3 (60 or 75mg/m² day or 20 or 25 mg/m² per day), repeated every 3 weeks, up to 3 cycles.
  Arms: Arm A
Drug: Ifosfamide or dacarbazine — A treatment cycle consists of 3 weeks. Treatment may continue up to 3 cycles. Ifosfamide will be administered from day 1 to day 3 (7,5-9 g/m² over 3 days with mesna and G-CSF) or dacarbazine (100 mg/m² 1 day or 450 mg/m² 2 days) as per local practices, repeated every 3 weeks, up to 3 cycles.
  Arms: Arm A
Drug: Doxorubicin — A treatment cycle consists of 3 weeks. Doxorubicin will be administered from day 1 to day 3 (60 or 75mg/m² day or 20 or 25 mg/m² per day), repeated every 3 weeks, up to 6 cycles.
  Arms: Arm B
Drug: Ifosfamide or dacarbazine — A treatment cycle consists of 3 weeks. Ifosfamide will be administered from day 1 to day 3 (7,5-9 g/m² over 3 days with mesna and G-CSF) or dacarbazine (100 mg/m² 1 day or 450 mg/m² 2 days) as per local practices, repeated every 3 weeks, up to 6 cycles.
  Arms: Arm B
Drug: At the discretion of the investigator — Drug at the discretion of the investigator.
  Arms: Prospective cohort

SUMMARY:
The primary objective of this trial is to investigate whether the addition of 3 additional neo-adjuvant cycles of chemotherapy (doxorubicin based chemotherapy) to standard management according to the ISG-STS 10-01 study (3 cycles of neoadjuvant doxorubicin based chemotherapy + surgery +/- radiotherapy) improves the outcome of high-risk CINSARC patients with resectable soft-tissue sarcoma (STS). Primary endpoint is metastatic progression-free survival (M-PFS, after 3 years of follow-up).

DETAILED DESCRIPTION:
For high-risk CINSARC patients, this is a multicenter randomized two-arm phase III trial, with a ratio 1:1:

* Arm A: standard management (3 cycles of neoadjuvant doxorubicin based chemotherapy + surgery +/- radiotherapy)
* Arm B: experimental arm (6 cycles of neoadjuvant doxorubicin based chemotherapy + surgery +/- radiotherapy)

For low-risk CINSARC patients, this a multicenter prospective cohort with treatment at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria :

1. Histologically confirmed soft-tissue sarcoma by the RRePS (Réseau de Référence en Pathologie des Sarcomes et des Viscères) network, as recommended by the French NCI,
2. Grade 2 or 3 according to the FNCLCC grading system,
3. Available archived tumour sample for research purpose,
4. Non-metastatic and resectable disease,
5. No prior treatment for the disease under study,
6. Age ≥ 18 years,
7. Life expectancy ≥ 3 months,
8. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1,
9. Patients must have measurable disease (lesion in previously irradiated field can be considered as measurable if progressive at inclusion according to RECIST 1.1) defined as per RECIST v1.1 with at least one lesion that can be measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm or ≥ 15mm in case of adenopathy,
10. Women of childbearing potential must have a negative serum pregnancy test before study entry. Both women and men must agree to use a medically acceptable method of contraception throughout the treatment period and for one year after discontinuation of treatment. Acceptable methods of contraception include intrauterine device (IUD), oral contraceptive, subdermal implant and double barrier. Subjects of childbearing potential are those who have not been surgically sterilized (e.g., vasectomy for males and hysterectomy for females) or have not been free from menses for ≥ 1 year,
11. Voluntarily signed and dated written informed consents prior to any study specific procedure,
12. Patients with a social security in compliance with the French law.

Exclusion Criteria :

1. Soft-tissue sarcoma with the following histological subtypes: well-differentiated liposarcoma, alveolar soft-part sarcoma, dermatofibrosarcoma protuberans, clearcell sarcoma, embryonal and alveolar rhabdomyosarcoma,
2. Prior or concurrent malignant disease diagnosed or treated in the last 2 years except for adequately treated in situ carcinoma of the cervix, basal or squamous skin cell carcinoma, or in situ transitional bladder cell carcinoma,
3. Any other contraindication to anthracycline, ifosfamide or dacarbazine chemotherapy,
4. Participation to a study involving a medical or therapeutic intervention in the last 28 days,
5. Known infection with HIV, hepatitis B, or hepatitis C,
6. Females who are pregnant or breast-feeding,
7. Other medical conditions may interfere with the conduct of the study and, in the judgment of the investigator, would make the patient inappropriate for entry into this study,
8. Individuals deprived of liberty or placed under legal guardianship,
9. Unwillingness or inability to comply with the study protocol for any reason.

Additional criteria for randomization :

1. High-risk CINSARC signature,
2. No more than two cycle of neo-adjuvant anthracycline-based chemotherapy before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Estimated)
Dates: Start 2019-02-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Metastasis progression-free survival in High-risk CINSARC patients | 3 years
  Metastasis progression-free survival (M-PFS) defined as the time interval between the date of randomization and the date of death or distant progression.

SECONDARY OUTCOMES:
Loco-regional relapse-free survival in High-risk CINSARC patients | 3 years
  Loco-regional relapse-free survival (LR-RFS) defined as the time interval between the randomization date and the date of death or loco-regional progression.
Progression-free survival in High-risk CINSARC patients | 3 years
  Progression-free survival (PFS) defined as the time interval between the randomization date and the date of death or progression (as per RECIST v1.1).
Overall survival in High-risk CINSARC patients | 3 years
  Overall survival (OS) defined as the time interval between the randomization date and the date of death.
Best overall response in High-risk CINSARC patients | Throughout the treatment period, an average of 6 months
  Best overall response under treatment as per RECIST v1.1.
Histological response in High-risk CINSARC patients | An average of 6 months
  Histological response defined as the proportion of recognizable cells on the tumor sample.
Safety profile in High-risk CINSARC patients | Throughout the treatment period, an average of 6 months
  Toxicity graded using the common toxicity criteria from the NCI v5.
Progression-free survival in Low-risk CINSARC patients | 3 years
  Progression-free survival defined as the time interval between the randomization date and the date of death or progression (as per RECIST v1.1).
Metastasis progression-free survival in Low-risk CINSARC patients | 3 years
  Metastasis progression-free survival defined as the time interval between the inclusion date and the date of death or distant progression.
Loco-regional progression-free survival in Low-risk CINSARC patients | 3 years
  Description of the treatment efficacy in terms of 3-years loco-regional progression-free survival defined as the time interval between the randomization date and the date of death or loco-regional progression.
Overall survival in Low-risk CINSARC patients | 3 years
  Overall survival defined as the time interval between the inclusion date and the date of death.

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Institut Bergonie, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - CHU Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Insitut du Cancer, Montpellier
  - Institut de Cancérologie de l'Ouest - Site René Gauducheau, Saint-Herblain
  - CHRU Strasbourg, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif